CLINICAL TRIAL: NCT02834780
Title: An Open-Label Multicenter Phase 1 Study to Evaluate the Safety, Pharmacokinetics and Pharmacodynamics of H3B-6527 in Subjects With Advanced Hepatocellular Carcinoma
Brief Title: Phase 1 Study to Evaluate the Safety, Pharmacokinetics and Pharmacodynamics of H3B-6527 in Participants With Advanced Hepatocellular Carcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H3 Biomedicine Inc. (Industry)
Collaborators: Eisai Inc. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H3B-6527-G000-101; 2016-001915-19 (EudraCT Number)
Record Dates: First submitted 2016-07-13; First posted 2016-07-15 (Estimated); Results first posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2021-07

CONDITIONS: Advanced Hepatocellular Carcinoma; Hepatocellular Carcinoma; Liver Cancer; Liver Neoplasms; Hepatic Cancer; Hepatic Carcinoma
Keywords: Advanced Hepatocellular Carcinoma; H3B-6527; Fibroblast growth factor receptor 4 (FGFR4); Fibroblast growth factor 19 (FGF19)
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — H3B-6527

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- H3B-6527 (escalation and expansion) (Experimental): Hepatocellular Carcinoma
  Interventions: Drug: H3B-6527

INTERVENTIONS:
Drug: H3B-6527 — H3B-6527 by mouth once or twice daily at specified doses.

SUMMARY:
The purpose of this study is to determine the maximum tolerated dose (MTD) and recommended Phase 2 dose (RP2D) of H3B-6527, and to assess the safety, tolerability and pharmacokinetics of H3B-6527.

ELIGIBILITY:
Inclusion criteria:

1. Participants with hepatocellular carcinoma.
2. Must have had at least one prior standard-of-care therapy, unless contraindicated.
3. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
4. Must be willing to undergo a biopsy up to 8 weeks before administration of H3B-6527 on Cycle 1 Day 1 for part 2 (dose expansion).
5. Adequate bone marrow and organ function.

Exclusion criteria:

1. Uncontrolled significant active infections, except hepatitis B virus (HBV) or hepatitis C virus (HCV).
2. Known human immunodeficiency virus infection.
3. Presence of gastric or esophageal varices requiring active treatment.
4. Previous treatment with a selective FGF19-FGFR4 targeted therapy.
5. Females of childbearing potential, or males who have not had a successful vasectomy, who are unable or unwilling to follow adequate contraceptive measures.
6. Hereditary problems of galactose intolerance, the Lapp lactase deficiency, or glucose-galactose malabsorption.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2016-12-28 (Actual); Primary Completion 2022-02-23 (Actual); Study Completion 2022-02-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (44):
- United States (15):
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - UC Irvine Medical Center, Orange, California
  - UCLA Medical Center, Santa Monica, California
  - Georgetown Unversity Lombardi Comprehensive Cancer Center, Washington D.C., District of Columbia
  - Northwestern Unversity, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - John theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Duke University Cancer Center, Durham, North Carolina
  - University of Cincinnati Cancer Institute, Cincinnati, Ohio
  - University of Pennsylsvania - Perelman Cancer Center for Advanced Medicine, Philadelphia, Pennsylvania
  - Simmons Comprehensive Cancer Center, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - McGuire VA Medical Center, Richmond, Virginia
- Belgium (2):
  - UCL Cliniques universitaires Saint-Luc, Woluwe-Saint-Lambert, Brussels Capital
  - Universitair Ziekenhuis Gent, Ghent
- Canada (2):
  - Cross Cancer Institute, Edmonton, Alberta
  - Jurvanski Cancer Center, Hamilton, Ontario
- France (4):
  - Institut Bergonié, Bordeaux
  - Centre Oscar Lambret, Lille
  - Hôpital Haut-Lévêque - CHU de Bordeaux, Pessac
  - Centre Eugène Marquis, Rennes
- Italy (3):
  - IRCCS Istituto Scientifico Romagnolo per lo studio e la cura dei tumori - U.O. di Oncologia Medica, Meldola
  - IRCCS Ospedale San Raffaele S.r.l. - PPDS, Milan
  - Azienda Ospedaliero Universitaria - Policlinico di Modena, Modena
- Russia (5):
  - Altay Regional Oncology Center, Barnaul, Altay, Re
  - Russian Oncology Research Center n a N N Blokhin, Moscow
  - Omsk Regional Oncology Center, Omsk
  - Railway Clinical Hospital JSC RZhD, Saint Petersburg
  - City Clinical Oncology Dispensary, Saint Petersburg
- National University Cancer Insitute, Singapore, Singapore
- Asan Medical Center, Seoul, South Korea
- Spain (8):
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - Clínica Universidad de Navarra, Pamplona, Navarre
  - Hospital Universitario de Badajoz, Badajoz
  - Hospital Universitario Vall d'Hebron, Barcelona
  - General Universitario Gregorio Maranon, Madrid
  - START Madrid FJD, Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario HM Sanchinarro, Madrid
  - Hospital Universitario Virgen del Rocio, Seville
- Taiwan (2):
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
- Sarah Cannon Research Institute UK - SCRI - PPDS, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 54 investigative sites in Belgium, Canada, France, Italy, Republic of Korea, Russian Federation, Singapore, Spain, Taiwan and the United States from 28 December 2016 to 23 February 2022.
Pre-assignment Details: A total of 304 participants were screened, of which 176 were screen failures and 128 were enrolled into two parts: Dose Escalation Phase (Part 1) and Dose Expansion Phase (Part 2) to receive study treatment.
Groups:
- Part 1, Dose Escalation Phase: H3B-6527 300 mg QD Fasted: Participants received H3B-6527 300 milligram (mg) capsule, orally, once daily (QD) in 21-days cycle in fasted state during treatment phase in dose escalation phase until disease progression, development of unacceptable toxicity, withdrawal of consent, or termination of the participants from the study by the Sponsor.
- Part 1, Dose Escalation Phase: H3B-6527 600 mg QD Fasted: Participants received H3B-6527 600 mg capsule, orally, QD in 21-days cycle in fasted state during treatment phase in dose escalation phase until disease progression, development of unacceptable toxicity, withdrawal of consent, or termination of the participants from the study by the Sponsor.
- Part 1, Dose Escalation Phase: H3B-6527 600 mg QD Fed: Participants received H3B-6527 600 mg capsule, orally, QD in 21-days cycle in fed state during treatment phase in dose escalation phase until disease progression, development of unacceptable toxicity, withdrawal of consent, or termination of the participants from the study by the Sponsor.
- Part 1, Dose Escalation Phase: H3B-6527 1000 mg QD Fasted: Participants received H3B-6527 1000 mg capsule, orally, QD in 21-days cycle in fasted state during treatment phase in dose escalation phase until disease progression, development of unacceptable toxicity, withdrawal of consent, or termination of the participants from the study by the Sponsor.
- Part 1, Dose Escalation Phase: H3B-6527 1000 mg QD Fed: Participants received H3B-6527 1000 mg capsule, orally, QD in 21-days cycle in fed state during treatment phase in dose escalation phase until disease progression, development of unacceptable toxicity, withdrawal of consent, or termination of the participants from the study by the Sponsor.
- Part 1, Dose Escalation Phase: H3B-6527 1400 mg QD Fasted: Participants received H3B-6527 1400 mg capsule, orally, QD in 21-days cycle in fasted state during treatment phase in dose escalation phase until disease progression, development of unacceptable toxicity, withdrawal of consent, or termination of the participants from the study by the Sponsor.
- Part 1, Dose Escalation Phase: H3B-6527 1400 mg QD Fed: Participants received H3B-6527 1400 mg capsule, orally, QD in 21-days cycle in fed state during treatment phase in dose escalation phase until disease progression, development of unacceptable toxicity, withdrawal of consent, or termination of the participants from the study by the Sponsor.
- Part 1, Dose Escalation Phase: H3B-6527 2000 mg QD Fed: Participants received H3B-6527 2000 mg capsule, orally, QD in 21-days cycle in fed state during treatment phase in dose escalation phase until disease progression, development of unacceptable toxicity, withdrawal of consent, or termination of the participants from the study by the Sponsor.
- Part 1, Dose Escalation Phase: H3B-6527 500 mg BID Fasted: Participants received H3B-6527 500 mg capsule, orally, twice a day (BID) in 21-days cycle in fasted state during treatment phase in dose escalation phase until disease progression, development of unacceptable toxicity, withdrawal of consent, or termination of the participants from the study by the Sponsor.
- Part 1, Dose Escalation Phase: H3B-6527 500 mg BID Fed: Participants received H3B-6527 500 mg capsule, orally, BID in 21-days cycle in fed state during treatment phase in dose escalation phase until disease progression, development of unacceptable toxicity, withdrawal of consent, or termination of the participants from the study by the Sponsor.
- Part 1, Dose Escalation Phase: H3B-6527 700 mg BID Fed: Participants received H3B-6527 700 mg capsule, orally, BID in 21-days cycle in fed state during treatment phase in dose escalation phase until disease progression, development of unacceptable toxicity, withdrawal of consent, or termination of the participants from the study by the Sponsor.
- Part 2, Dose Expansion Phase: H3B-6527 1000 mg QD: Participants received H3B-6527 1000 mg capsule, orally, QD in 21-days cycle either in fasted or fed state during treatment phase in dose expansion phase until disease progression, development of unacceptable toxicity, withdrawal of consent, or termination of the participants from the study by the Sponsor.
- Part 2, Dose Expansion Phase: H3B-6527 500 mg BID Fed: Participants received H3B-6527 500 mg capsule, orally, BID in 21-days cycle in fed state during treatment phase in dose expansion phase until disease progression, development of unacceptable toxicity, withdrawal of consent, or termination of the participants from the study by the Sponsor.
Period: Overall Study
Arm/Group | Part 1, Dose Escalation Phase: H3B-6527 300 mg QD Fasted | Part 1, Dose Escalation Phase: H3B-6527 600 mg QD Fasted | Part 1, Dose Escalation Phase: H3B-6527 600 mg QD Fed | Part 1, Dose Escalation Phase: H3B-6527 1000 mg QD Fasted | Part 1, Dose Escalation Phase: H3B-6527 1000 mg QD Fed | Part 1, Dose Escalation Phase: H3B-6527 1400 mg QD Fasted | Part 1, Dose Escalation Phase: H3B-6527 1400 mg QD Fed | Part 1, Dose Escalation Phase: H3B-6527 2000 mg QD Fed | Part 1, Dose Escalation Phase: H3B-6527 500 mg BID Fasted | Part 1, Dose Escalation Phase: H3B-6527 500 mg BID Fed | Part 1, Dose Escalation Phase: H3B-6527 700 mg BID Fed | Part 2, Dose Expansion Phase: H3B-6527 1000 mg QD | Part 2, Dose Expansion Phase: H3B-6527 500 mg BID Fed
Started | 3 | 3 | 4 | 10 | 3 | 7 | 4 | 7 | 3 | 10 | 5 | 29 | 40
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 3 | 4 | 10 | 3 | 7 | 4 | 7 | 3 | 10 | 5 | 29 | 40
Not completed — Disease Progression -Radiologically Confirmed | 1 | 3 | 2 | 7 | 1 | 6 | 2 | 4 | 3 | 6 | 3 | 24 | 32
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 2 | 0 | 3 | 2
Not completed — Disease Progression - Clinically Confirmed | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 2 | 0 | 2 | 1 | 2 | 5
Not completed — Other | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set included all participants who received at least 1 dose of the study drug.
Groups:
- Part 1, Dose Escalation Phase: H3B-6527 300 mg QD Fasted: Participants received H3B-6527 300 mg capsule, orally, QD in 21-days cycle in fasted state during treatment phase in dose escalation phase until disease progression, development of unacceptable toxicity, withdrawal of consent, or termination of the participants from the study by the Sponsor.
- Part 1, Dose Escalation Phase: H3B-6527 500 mg BID Fasted: Participants received H3B-6527 500 mg capsule, orally, BID in 21-days cycle in fasted state during treatment phase in dose escalation phase until disease progression, development of unacceptable toxicity, withdrawal of consent, or termination of the participants from the study by the Sponsor.
- Total: Total of all reporting groups
Arm/Group | Part 1, Dose Escalation Phase: H3B-6527 300 mg QD Fasted | Part 1, Dose Escalation Phase: H3B-6527 600 mg QD Fasted | Part 1, Dose Escalation Phase: H3B-6527 600 mg QD Fed | Part 1, Dose Escalation Phase: H3B-6527 1000 mg QD Fasted | Part 1, Dose Escalation Phase: H3B-6527 1000 mg QD Fed | Part 1, Dose Escalation Phase: H3B-6527 1400 mg QD Fasted | Part 1, Dose Escalation Phase: H3B-6527 1400 mg QD Fed | Part 1, Dose Escalation Phase: H3B-6527 2000 mg QD Fed | Part 1, Dose Escalation Phase: H3B-6527 500 mg BID Fasted | Part 1, Dose Escalation Phase: H3B-6527 500 mg BID Fed | Part 1, Dose Escalation Phase: H3B-6527 700 mg BID Fed | Part 2, Dose Expansion Phase: H3B-6527 1000 mg QD | Part 2, Dose Expansion Phase: H3B-6527 500 mg BID Fed | Total
Number analyzed (Participants) | 3 | 3 | 4 | 10 | 3 | 7 | 4 | 7 | 3 | 10 | 5 | 29 | 40 | 128
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.0 (7.00) | 72.7 (4.73) | 68.5 (9.75) | 67.1 (8.01) | 68.7 (6.51) | 59.3 (12.22) | 60.3 (7.14) | 62.1 (7.52) | 68.7 (4.04) | 62.0 (16.51) | 65.6 (9.91) | 61.4 (10.67) | 64.3 (10.58) | 63.6 (10.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 2 | 2 | 0 | 3 | 2 | 3 | 1 | 3 | 2 | 7 | 12 | 37
  Male | 3 | 3 | 2 | 8 | 3 | 4 | 2 | 4 | 2 | 7 | 3 | 22 | 28 | 91
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 5
  Not Hispanic or Latino | 3 | 3 | 4 | 9 | 3 | 7 | 4 | 6 | 3 | 9 | 5 | 27 | 28 | 111
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 10 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 1 | 1 | 1 | 2 | 2 | 0 | 0 | 5 | 2 | 8 | 7 | 30
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 5
  White | 2 | 3 | 2 | 9 | 1 | 4 | 1 | 7 | 3 | 4 | 3 | 20 | 22 | 81
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 10 | 11

OUTCOME MEASURES:

1. Primary Outcome: Part 1, Dose Escalation Phase: Number of Participants With Dose-limiting Toxicities (DLTs) Based on National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03
Description: DLTs were defined as any of the following toxicities: Hematology, gastrointestinal, renal, hepatic or nonhematologic toxicities occurring during Cycle 1 in Dose Escalation Phase only and judged by the investigator as related to study drug. This included any Grade 4: neutropenia that does not resolve to Grade less than or equal to (<=) 2 within 7 days, thrombocytopenia, anemia of any duration, diarrhea and/or vomiting irrespective of prophylaxis or appropriate treatment; Grade 3: thrombocytopenia requiring transfusion, thrombocytopenia and clinically significant bleeding, anemia if transfused or if lasting for more than 7 days, nausea, vomiting and/or diarrhea lasting more than 72 hours despite the use of optimal anti-emetic/antidiarrheal treatment, bilirubin, fatigue lasting less than 1 week, elevations in biochemistry laboratory values without associated clinical symptoms that last for <=7 days; Grade greater than or equal to (>=) 3 serum creatinine.
Time Frame: Cycle 1 (Cycle length = 21 days)
Population: DLT analysis set included all participants in Dose Escalation phase (Part 1) who must have completed safety assessments through pre-dose on Cycle 2 Day 1 and must have received at least 17 of 21 (approximately 80 percent [%]) study days within Cycle 1, unless due to a DLT. This outcome measure was planned to be analyzed for Part 1 only.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1, Dose Escalation Phase: H3B-6527 300 mg QD Fasted | Part 1, Dose Escalation Phase: H3B-6527 600 mg QD Fasted | Part 1, Dose Escalation Phase: H3B-6527 600 mg QD Fed | Part 1, Dose Escalation Phase: H3B-6527 1000 mg QD Fasted | Part 1, Dose Escalation Phase: H3B-6527 1000 mg QD Fed | Part 1, Dose Escalation Phase: H3B-6527 1400 mg QD Fasted | Part 1, Dose Escalation Phase: H3B-6527 1400 mg QD Fed | Part 1, Dose Escalation Phase: H3B-6527 2000 mg QD Fed | Part 1, Dose Escalation Phase: H3B-6527 500 mg BID Fasted | Part 1, Dose Escalation Phase: H3B-6527 500 mg BID Fed | Part 1, Dose Escalation Phase: H3B-6527 700 mg BID Fed
Number analyzed (Participants) | 3 | 3 | 4 | 10 | 3 | 6 | 3 | 7 | 3 | 9 | 4
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: A TEAE was defined as an adverse event (AE) that emerges during treatment, having been absent at pretreatment (Baseline) or reemerges during treatment, having been present at pretreatment (Baseline) but stopped before treatment, or worsens in severity during treatment relative to the pretreatment state, when the AE was continuous. An SAE was any untoward medical occurrence that at any dose: Resulted in death, was life-threatening (that is, the participant was at immediate risk of death from the AE as it occurred; this does not include an event that, had it occurred in a more severe form or was allowed to continue, might have caused death), required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect (in the child of a participant who was exposed to the study drug).
Time Frame: From the first dose of study drug up to approximately 36.7 months
Population: Safety analysis set included all participants who received at least 1 dose of the study drug. This outcome measure was planned to be analyzed for Part 1 and Part 2.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1, Dose Escalation Phase: H3B-6527 300 mg QD Fasted | Part 1, Dose Escalation Phase: H3B-6527 600 mg QD Fasted | Part 1, Dose Escalation Phase: H3B-6527 600 mg QD Fed | Part 1, Dose Escalation Phase: H3B-6527 1000 mg QD Fasted | Part 1, Dose Escalation Phase: H3B-6527 1000 mg QD Fed | Part 1, Dose Escalation Phase: H3B-6527 1400 mg QD Fasted | Part 1, Dose Escalation Phase: H3B-6527 1400 mg QD Fed | Part 1, Dose Escalation Phase: H3B-6527 2000 mg QD Fed | Part 1, Dose Escalation Phase: H3B-6527 500 mg BID Fasted | Part 1, Dose Escalation Phase: H3B-6527 500 mg BID Fed | Part 1, Dose Escalation Phase: H3B-6527 700 mg BID Fed | Part 2, Dose Expansion Phase: H3B-6527 1000 mg QD | Part 2, Dose Expansion Phase: H3B-6527 500 mg BID Fed
Number analyzed (Participants) | 3 | 3 | 4 | 10 | 3 | 7 | 4 | 7 | 3 | 10 | 5 | 29 | 40
Participants
  Participants with TEAEs | 3 | 3 | 4 | 10 | 3 | 7 | 4 | 7 | 3 | 9 | 5 | 28 | 40
  Participants with SAEs | 0 | 0 | 1 | 1 | 1 | 4 | 1 | 2 | 2 | 3 | 1 | 11 | 17

3. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time 0 Through the Last Measurable Point (AUC0-t) of H3B-6527
Time Frame: Part 1, Cycle 1 Day 1 and Day 8: 0-24 hours post-dose (for QD dosing) and 0-10 hours post-dose (for BID dosing); Part 2, Cycle 1 Day 8: 0-24 hours post-dose (for QD dosing) and 0-10 hours post-dose (for BID dosing) (Cycle 1 length = 21 days)
Population: Pharmacokinetic (PK) analysis set: Participants who received at least 1 dose of study drug and had at least 1 evaluable plasma concentration. 'Overall Number of participants analyzed' signifies those who were evaluable for this outcome measure; 'Number analyzed' signifies participants who were evaluable at given timepoints. As planned, PK data was collected and reported together due to same dose and food conditions in Part 1 and 2 for H3B-6527 1000 mg (QD fed and fasted) and 500 mg (BID fed).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*h/mL)
Groups:
- Parts 1 and 2, Dose Escalation + Expansion Phase: H3B-6527 1000 mg QD Fasted: Participants received H3B-6527 1000 mg capsule, orally, QD in 21-days cycle in fasted state during treatment phase of dose escalation and expansion phases until disease progression, development of unacceptable toxicity, withdrawal of consent, or termination of the study by the Sponsor.
- Parts 1 and 2, Dose Escalation + Expansion Phase: H3B-6527 1000 mg QD Fed: Participants received H3B-6527 1000 mg capsule, orally, QD in 21-days cycle in fed state during treatment phase of dose escalation and expansion phases until disease progression, development of unacceptable toxicity, withdrawal of consent, or termination of the study by the Sponsor.
- Parts 1 and 2, Dose Escalation + Expansion Phase: H3B-6527 500 mg BID Fed: Participants received H3B-6527 500 mg capsules, orally, BID in 21-days cycle in fed state during treatment phase of dose escalation and expansion phases until disease progression, development of unacceptable toxicity, withdrawal of consent, or termination of the study by the Sponsor.
Arm/Group | Part 1, Dose Escalation Phase: H3B-6527 300 mg QD Fasted | Part 1, Dose Escalation Phase: H3B-6527 600 mg QD Fasted | Part 1, Dose Escalation Phase: H3B-6527 600 mg QD Fed | Parts 1 and 2, Dose Escalation + Expansion Phase: H3B-6527 1000 mg QD Fasted | Parts 1 and 2, Dose Escalation + Expansion Phase: H3B-6527 1000 mg QD Fed | Part 1, Dose Escalation Phase: H3B-6527 1400 mg QD Fasted | Part 1, Dose Escalation Phase: H3B-6527 1400 mg QD Fed | Part 1, Dose Escalation Phase: H3B-6527 2000 mg QD Fed | Part 1, Dose Escalation Phase: H3B-6527 500 mg BID Fasted | Parts 1 and 2, Dose Escalation + Expansion Phase: H3B-6527 500 mg BID Fed | Part 1, Dose Escalation Phase: H3B-6527 700 mg BID Fed
Number analyzed (Participants) | 3 | 3 | 4 | 32 | 7 | 7 | 4 | 7 | 3 | 45 | 5
nanogram*hour per milliliter (ng*h/mL)
  Cycle 1 Day 1: number analyzed (Participants) | 3 | 3 | 3 | 9 | 3 | 7 | 4 | 7 | 3 | 10 | 5
  Cycle 1 Day 1 | 68.9 (57.5) | 173 (1891.9) | 1631 (271.8) | 850 (531.5) | 1115 (909.7) | 400 (187.5) | 5671 (98.7) | 2748 (66.3) | 462 (137.0) | 752 (204.3) | 576 (482.6)
  Cycle 1 Day 8 | 50.8 (47.5) | 636 (39.4) | 484 (3217.3) | 784 (431.8) | 798 (337.8) | 1244 (827.7) | 5447 (74.9) | 1838 (179.3) | 1056 (36.9) | 809 (237.3) | 622 (351.1)

4. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of H3B-6527
Time Frame: as for outcome 3
Population: PK analysis set: Participants who received at least 1 dose of study drug and had at least 1 evaluable plasma concentration. 'Overall Number of participants analyzed' signifies those who were evaluable for this outcome measure; 'Number analyzed' signifies participants who were evaluable at given timepoints. As planned, PK data was collected and reported together due to same dose and food conditions in Part 1 and 2 for H3B-6527 1000 mg (QD fed and fasted) and 500 mg (BID fed).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Part 1, Dose Escalation Phase: H3B-6527 300 mg QD Fasted | Part 1, Dose Escalation Phase: H3B-6527 600 mg QD Fasted | Part 1, Dose Escalation Phase: H3B-6527 600 mg QD Fed | Parts 1 and 2, Dose Escalation + Expansion Phase: H3B-6527 1000 mg QD Fasted | Parts 1 and 2, Dose Escalation + Expansion Phase: H3B-6527 1000 mg QD Fed | Part 1, Dose Escalation Phase: H3B-6527 1400 mg QD Fasted | Part 1, Dose Escalation Phase: H3B-6527 1400 mg QD Fed | Part 1, Dose Escalation Phase: H3B-6527 2000 mg QD Fed | Part 1, Dose Escalation Phase: H3B-6527 500 mg BID Fasted | Parts 1 and 2, Dose Escalation + Expansion Phase: H3B-6527 500 mg BID Fed | Part 1, Dose Escalation Phase: H3B-6527 700 mg BID Fed
Number analyzed (Participants) | 3 | 3 | 4 | 32 | 7 | 7 | 4 | 7 | 3 | 45 | 5
nanogram per milliliter (ng/mL)
  Cycle 1 Day 1: number analyzed (Participants) | 3 | 3 | 3 | 9 | 3 | 7 | 4 | 7 | 3 | 10 | 5
  Cycle 1 Day 1 | 20.3 (64.1) | 74.5 (1389.4) | 395 (133.7) | 225 (470.2) | 182 (494.6) | 136 (429.4) | 904 (34.2) | 540 (79.9) | 124 (159.1) | 255 (251.6) | 163 (303.2)
  Cycle 1 Day 8 | 10.8 (90.6) | 194 (45.6) | 99.6 (5300.4) | 187 (339.1) | 177 (370.3) | 362 (898.5) | 827 (40.6) | 502 (95.2) | 251 (46.5) | 211 (237.2) | 167 (202.7)

5. Secondary Outcome: Time of Maximum Observed Plasma Concentration (Tmax) of H3B-6527
Time Frame: as for outcome 3
Population: as for outcome 4
Measure: Median (Full Range); unit: hours
Arm/Group | Part 1, Dose Escalation Phase: H3B-6527 300 mg QD Fasted | Part 1, Dose Escalation Phase: H3B-6527 600 mg QD Fasted | Part 1, Dose Escalation Phase: H3B-6527 600 mg QD Fed | Parts 1 and 2, Dose Escalation + Expansion Phase: H3B-6527 1000 mg QD Fasted | Parts 1 and 2, Dose Escalation + Expansion Phase: H3B-6527 1000 mg QD Fed | Part 1, Dose Escalation Phase: H3B-6527 1400 mg QD Fasted | Part 1, Dose Escalation Phase: H3B-6527 1400 mg QD Fed | Part 1, Dose Escalation Phase: H3B-6527 2000 mg QD Fed | Part 1, Dose Escalation Phase: H3B-6527 500 mg BID Fasted | Parts 1 and 2, Dose Escalation + Expansion Phase: H3B-6527 500 mg BID Fed | Part 1, Dose Escalation Phase: H3B-6527 700 mg BID Fed
Number analyzed (Participants) | 3 | 3 | 4 | 32 | 7 | 7 | 4 | 7 | 3 | 45 | 5
hours
  Cycle 1 Day 1: number analyzed (Participants) | 3 | 3 | 3 | 9 | 3 | 7 | 4 | 7 | 3 | 10 | 5
  Cycle 1 Day 1 | 2.00 [2.00 to 4.00] | 1.00 [0.50 to 2.00] | 4.00 [1.00 to 4.07] | 2.02 [1.00 to 8.12] | 6.00 [4.10 to 6.00] | 1.00 [0.63 to 4.15] | 5.00 [2.00 to 8.00] | 2.100 [1.00 to 4.92] | 2.12 [2.00 to 4.57] | 4.02 [0.57 to 10.00] | 2.02 [0.50 to 6.12]
  Cycle 1 Day 8 | 4.00 [2.07 to 4.00] | 0.52 [0.50 to 2.00] | 4.52 [0.53 to 6.00] | 2.00 [0.33 to 10.00] | 2.00 [1.00 to 4.33] | 2.10 [1.00 to 4.13] | 5.86 [2.00 to 6.22] | 4.00 [1.00 to 8.42] | 4.00 [2.10 to 4.17] | 4.00 [0.00 to 10.00] | 4.12 [0.50 to 10.00]

6. Secondary Outcome: Part 2, Dose Expansion Phase: Objective Response Rate (ORR) Based on Modified Response Evaluation Criteria in Solid Tumors (mRECIST) v1.1
Description: ORR was defined as the percentage of participants achieving a best overall confirmed response of partial response (PR) or complete response (CR) (PR + CR), from the first dose date until disease progression/recurrence. Responses (PR or CR) were confirmed no less than 4 weeks after the initial response. CR was defined as the disappearance of all target lesions and non-target lesions. Any pathological lymph nodes (target or non-target) had to be reduced in the short axis to less than 10 millimeter (mm). PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters. The tumor assessment was done using number of lesions based on modified RECIST v1.1 for assessing tumor burden up to 10 target lesions with up to 5 target lesions per organ.
Time Frame: From the first dose date until disease progression/recurrence or up to approximately 36.7 months
Population: Full analysis set included all participants who received at least 1 dose of the study drug. Here, "overall number of participants analyzed" signifies participants who were evaluable for this outcome measure. This outcome measure was planned to be analyzed for Part 2 only.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Part 2, Dose Expansion Phase: H3B-6527 1000 mg QD: Participants with hepatocellular carcinoma (HCC) received H3B-6527 1000 mg capsule, orally, QD in 21-days cycle either in fasted or fed state during treatment phase in dose expansion phase until disease progression, development of unacceptable toxicity, withdrawal of consent, or termination of the participants from the study by the Sponsor.
- Part 2, Dose Expansion Phase: H3B-6527 500 mg BID Fed: Participants with HCC received H3B-6527 500 mg capsule, orally, BID in 21-days cycle in fed state during treatment phase in dose expansion phase until disease progression, development of unacceptable toxicity, withdrawal of consent, or termination of the participants from the study by the Sponsor.
Arm/Group | Part 2, Dose Expansion Phase: H3B-6527 1000 mg QD | Part 2, Dose Expansion Phase: H3B-6527 500 mg BID Fed
Number analyzed (Participants) | 18 | 32
percentage of participants | 5.6 [0.1 to 27.3] | 0.0 [0.0 to 10.9]

7. Secondary Outcome: Part 2, Dose Expansion Phase: Duration of Response (DOR) Based on Modified Response Evaluation Criteria in Solid Tumors (mRECIST) v1.1
Description: DOR was defined as the time from the date of first documented CR or PR based on modified RECIST v1.1 until the first documentation of disease progression (PD) as determined by the investigator or death, whichever comes first. CR was defined as the disappearance of all target lesions and non-target lesions. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters. PD was defined as at least a 20% increase in the sum of long diameter (LD) of target and non-target lesions as compared with the smallest sum of LD and the increase of LD was at least 5 mm (including new lesions).
Time Frame: From the date of first documented CR or PR up to approximately 36.7 months
Population: Full analysis set included all participants who received at least 1 dose of the study drug. Here, overall number of participants analyzed "N" included the participants who had CR or PR. This outcome measure was planned to be analyzed for Part 2 only.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Part 2, Dose Expansion Phase: H3B-6527 1000 mg QD: Participants with HCC received H3B-6527 1000 mg capsule, orally, QD in 21-days cycle either in fasted or fed state during treatment phase in dose expansion phase until disease progression, development of unacceptable toxicity, withdrawal of consent, or termination of the participants from the study by the Sponsor.
Arm/Group | Part 2, Dose Expansion Phase: H3B-6527 1000 mg QD | Part 2, Dose Expansion Phase: H3B-6527 500 mg BID Fed
Number analyzed (Participants) | 1 | 0
months | NA [NA to NA] — The DOR could not be evaluated due to the small number of responders participants. |

8. Secondary Outcome: Part 2, Dose Expansion Phase: Progression-free Survival (PFS) Based on Modified Response Evaluation Criteria in Solid Tumors (mRECIST) v1.1
Description: PFS was defined as the time from the first dose date to the date of the first documentation of PD as determined by the investigator or death (whichever occurs first). PD was defined as at least a 20% increase in the sum of LD of target and non-target lesions as compared with the smallest sum of LD and the increase of LD was at least 5 mm (including new lesions).
Time Frame: From the first dose date to the date of the first documentation of PD as determined by the investigator or death (whichever occurs first) up to approximately 36.7 months
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part 2, Dose Expansion Phase: H3B-6527 1000 mg QD | Part 2, Dose Expansion Phase: H3B-6527 500 mg BID Fed
Number analyzed (Participants) | 18 | 32
months | 2.6 [1.3 to 5.5] | 3.0 [1.5 to 4.1]

9. Secondary Outcome: Part 2, Dose Expansion Phase: Overall Survival (OS)
Description: OS was defined as the time from the first dose date to the date of death. OS was assessed using Kaplan-Meier method. The time of death was censored for participants who were without death information at the time of OS analysis.
Time Frame: From the date of first dose of study drug until date of death from any cause (up to approximately 36.7 months)
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part 2, Dose Expansion Phase: H3B-6527 1000 mg QD | Part 2, Dose Expansion Phase: H3B-6527 500 mg BID Fed
Number analyzed (Participants) | 18 | 32
months | 9.5 [2.3 to 24.4] | 7.7 [4.7 to 11.3]

10. Secondary Outcome: Part 2, Dose Expansion Phase: Time to Response (TTR) Based on Modified Response Evaluation Criteria in Solid Tumors (mRECIST) v1.1
Description: TTR was defined as the time from the first dose date to the date of first documented CR/PR. CR was defined as the disappearance of all target lesions and non-target lesions. Any pathological lymph nodes (target or non-target) had to be reduced in the short axis to less than 10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters.
Time Frame: From date of first dose of study drug until CR or PR (up to approximately 36.7 months)
Population: Full analysis set included all participants who received at least 1 dose of the study drug. Here, "overall number of participants analyzed" signifies participants who had CR or PR. This outcome measure was planned to be analyzed for Part 2 only.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part 2, Dose Expansion Phase: H3B-6527 1000 mg QD | Part 2, Dose Expansion Phase: H3B-6527 500 mg BID Fed
Number analyzed (Participants) | 1 | 0
months | NA [NA to NA] — The TTR could not be evaluated due to the small number of responders participants. |

11. Primary Outcome: Number of Participants With Clinically Significant Change From Baseline in Laboratory Parameters
Description: Laboratory assessment included hematology, coagulation, clinical chemistry, and urinalysis parameters.
Time Frame: From baseline up to approximately 36.7 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1, Dose Escalation Phase: H3B-6527 300 mg QD Fasted | Part 1, Dose Escalation Phase: H3B-6527 600 mg QD Fasted | Part 1, Dose Escalation Phase: H3B-6527 600 mg QD Fed | Part 1, Dose Escalation Phase: H3B-6527 1000 mg QD Fasted | Part 1, Dose Escalation Phase: H3B-6527 1000 mg QD Fed | Part 1, Dose Escalation Phase: H3B-6527 1400 mg QD Fasted | Part 1, Dose Escalation Phase: H3B-6527 1400 mg QD Fed | Part 1, Dose Escalation Phase: H3B-6527 2000 mg QD Fed | Part 1, Dose Escalation Phase: H3B-6527 500 mg BID Fasted | Part 1, Dose Escalation Phase: H3B-6527 500 mg BID Fed | Part 1, Dose Escalation Phase: H3B-6527 700 mg BID Fed | Part 2, Dose Expansion Phase: H3B-6527 1000 mg QD | Part 2, Dose Expansion Phase: H3B-6527 500 mg BID Fed
Number analyzed (Participants) | 3 | 3 | 4 | 10 | 3 | 7 | 4 | 7 | 3 | 10 | 5 | 29 | 40
Participants
  Hematology | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Clinical Chemistry | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Urinalysis | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Coagulation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

12. Primary Outcome: Number of Participants With Clinically Significant Change From Baseline in Electrocardiogram (ECG) Parameters
Time Frame: From baseline up to approximately 36.7 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1, Dose Escalation Phase: H3B-6527 300 mg QD Fasted | Part 1, Dose Escalation Phase: H3B-6527 600 mg QD Fasted | Part 1, Dose Escalation Phase: H3B-6527 600 mg QD Fed | Part 1, Dose Escalation Phase: H3B-6527 1000 mg QD Fasted | Part 1, Dose Escalation Phase: H3B-6527 1000 mg QD Fed | Part 1, Dose Escalation Phase: H3B-6527 1400 mg QD Fasted | Part 1, Dose Escalation Phase: H3B-6527 1400 mg QD Fed | Part 1, Dose Escalation Phase: H3B-6527 2000 mg QD Fed | Part 1, Dose Escalation Phase: H3B-6527 500 mg BID Fasted | Part 1, Dose Escalation Phase: H3B-6527 500 mg BID Fed | Part 1, Dose Escalation Phase: H3B-6527 700 mg BID Fed | Part 2, Dose Expansion Phase: H3B-6527 1000 mg QD | Part 2, Dose Expansion Phase: H3B-6527 500 mg BID Fed
Number analyzed (Participants) | 3 | 3 | 4 | 10 | 3 | 7 | 4 | 7 | 3 | 10 | 5 | 29 | 40
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

13. Primary Outcome: Number of Participants With Clinically Significant Change From Baseline in Vital Sign Parameters
Time Frame: From baseline up to approximately 36.7 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1, Dose Escalation Phase: H3B-6527 300 mg QD Fasted | Part 1, Dose Escalation Phase: H3B-6527 600 mg QD Fasted | Part 1, Dose Escalation Phase: H3B-6527 600 mg QD Fed | Part 1, Dose Escalation Phase: H3B-6527 1000 mg QD Fasted | Part 1, Dose Escalation Phase: H3B-6527 1000 mg QD Fed | Part 1, Dose Escalation Phase: H3B-6527 1400 mg QD Fasted | Part 1, Dose Escalation Phase: H3B-6527 1400 mg QD Fed | Part 1, Dose Escalation Phase: H3B-6527 2000 mg QD Fed | Part 1, Dose Escalation Phase: H3B-6527 500 mg BID Fasted | Part 1, Dose Escalation Phase: H3B-6527 500 mg BID Fed | Part 1, Dose Escalation Phase: H3B-6527 700 mg BID Fed | Part 2, Dose Expansion Phase: H3B-6527 1000 mg QD | Part 2, Dose Expansion Phase: H3B-6527 500 mg BID Fed
Number analyzed (Participants) | 3 | 3 | 4 | 10 | 3 | 7 | 4 | 7 | 3 | 10 | 5 | 29 | 40
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From the first dose of study drug up to approximately 36.7 months
Arm/Group | Part 1, Dose Escalation Phase: H3B-6527 300 mg QD Fasted | Part 1, Dose Escalation Phase: H3B-6527 600 mg QD Fasted | Part 1, Dose Escalation Phase: H3B-6527 600 mg QD Fed | Part 1, Dose Escalation Phase: H3B-6527 1000 mg QD Fasted | Part 1, Dose Escalation Phase: H3B-6527 1000 mg QD Fed | Part 1, Dose Escalation Phase: H3B-6527 1400 mg QD Fasted | Part 1, Dose Escalation Phase: H3B-6527 1400 mg QD Fed | Part 1, Dose Escalation Phase: H3B-6527 2000 mg QD Fed | Part 1, Dose Escalation Phase: H3B-6527 500 mg BID Fasted | Part 1, Dose Escalation Phase: H3B-6527 500 mg BID Fed | Part 1, Dose Escalation Phase: H3B-6527 700 mg BID Fed | Part 2, Dose Expansion Phase: H3B-6527 1000 mg QD | Part 2, Dose Expansion Phase: H3B-6527 500 mg BID Fed
All-Cause Mortality (participants affected / at risk) | 1/3 | 3/3 | 2/4 | 6/10 | 2/3 | 7/7 | 3/4 | 1/7 | 3/3 | 6/10 | 4/5 | 19/29 | 31/40
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 1/4 | 1/10 | 1/3 | 4/7 | 1/4 | 2/7 | 2/3 | 3/10 | 1/5 | 11/29 | 17/40
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 4/4 | 10/10 | 3/3 | 7/7 | 4/4 | 7/7 | 3/3 | 9/10 | 5/5 | 28/29 | 39/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1, Dose Escalation Phase: H3B-6527 300 mg QD Fasted (N=3) | Part 1, Dose Escalation Phase: H3B-6527 600 mg QD Fasted (N=3) | Part 1, Dose Escalation Phase: H3B-6527 600 mg QD Fed (N=4) | Part 1, Dose Escalation Phase: H3B-6527 1000 mg QD Fasted (N=10) | Part 1, Dose Escalation Phase: H3B-6527 1000 mg QD Fed (N=3) | Part 1, Dose Escalation Phase: H3B-6527 1400 mg QD Fasted (N=7) | Part 1, Dose Escalation Phase: H3B-6527 1400 mg QD Fed (N=4) | Part 1, Dose Escalation Phase: H3B-6527 2000 mg QD Fed (N=7) | Part 1, Dose Escalation Phase: H3B-6527 500 mg BID Fasted (N=3) | Part 1, Dose Escalation Phase: H3B-6527 500 mg BID Fed (N=10) | Part 1, Dose Escalation Phase: H3B-6527 700 mg BID Fed (N=5) | Part 2, Dose Expansion Phase: H3B-6527 1000 mg QD (N=29) | Part 2, Dose Expansion Phase: H3B-6527 500 mg BID Fed (N=40)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hepatic haemorrhage (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Hepatic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Tumour rupture (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Immune thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Varices oesophageal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Incarcerated hernia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Jaundice (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1, Dose Escalation Phase: H3B-6527 300 mg QD Fasted (N=3) | Part 1, Dose Escalation Phase: H3B-6527 600 mg QD Fasted (N=3) | Part 1, Dose Escalation Phase: H3B-6527 600 mg QD Fed (N=4) | Part 1, Dose Escalation Phase: H3B-6527 1000 mg QD Fasted (N=10) | Part 1, Dose Escalation Phase: H3B-6527 1000 mg QD Fed (N=3) | Part 1, Dose Escalation Phase: H3B-6527 1400 mg QD Fasted (N=7) | Part 1, Dose Escalation Phase: H3B-6527 1400 mg QD Fed (N=4) | Part 1, Dose Escalation Phase: H3B-6527 2000 mg QD Fed (N=7) | Part 1, Dose Escalation Phase: H3B-6527 500 mg BID Fasted (N=3) | Part 1, Dose Escalation Phase: H3B-6527 500 mg BID Fed (N=10) | Part 1, Dose Escalation Phase: H3B-6527 700 mg BID Fed (N=5) | Part 2, Dose Expansion Phase: H3B-6527 1000 mg QD (N=29) | Part 2, Dose Expansion Phase: H3B-6527 500 mg BID Fed (N=40)
Anaemia (Blood and lymphatic system disorders) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 4 (7)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (7)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Supraventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deafness (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blepharitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cataract nuclear (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chalazion (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Corneal thinning (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Keratitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Open angle glaucoma (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periorbital oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinal haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Swelling of eyelid (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 2 (3) | 1 (1) | 2 (4) | 1 (1) | 0 (0) | 1 (1) | 5 (6) | 9 (9)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (4) | 3 (3)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 4 (7) | 3 (6)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (4) | 3 (4) | 7 (13) | 2 (3) | 4 (6) | 2 (2) | 4 (10) | 2 (5) | 6 (6) | 3 (3) | 10 (22) | 27 (45)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Faeces discoloured (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (4) | 4 (7) | 1 (1) | 4 (5) | 2 (2) | 4 (7) | 0 (0) | 2 (2) | 0 (0) | 6 (7) | 8 (10)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 4 (6) | 1 (1) | 3 (11) | 0 (0) | 0 (0) | 1 (1) | 5 (6) | 4 (9)
Paraesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 5 (9) | 6 (8)
Cyst (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 2 (3) | 2 (2) | 4 (8) | 1 (1) | 0 (0) | 2 (2) | 3 (5) | 9 (14)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (7) | 5 (6)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 2 (2)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatomegaly (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatorenal syndrome (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peritonitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Breast injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Intentional overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Activated partial thromboplastin time shortened (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (4) | 0 (0) | 2 (5) | 0 (0) | 2 (2) | 0 (0) | 4 (6) | 0 (0) | 2 (2) | 2 (3) | 0 (0) | 10 (24)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 2 (4) | 0 (0) | 2 (15) | 0 (0) | 2 (2) | 2 (3) | 4 (10) | 0 (0) | 1 (1) | 2 (3) | 2 (7) | 14 (34)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 3 (7) | 0 (0) | 0 (0) | 1 (4) | 2 (2) | 1 (11)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (5) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 9 (21)
Blood cholesterol increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (8) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (3) | 1 (2) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood potassium increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood uric acid increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood urine present (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Human metapneumovirus test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (4) | 4 (4)
Total bile acids increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Transaminases increased (Investigations) | 1 (3) | 0 (0) | 0 (0) | 2 (9) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 3 (3)
Waist circumference increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (8)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (2) | 4 (7) | 11 (13)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (24) | 0 (0) | 0 (0) | 0 (0) | 2 (15) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (6)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (3)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 4 (4)
Coccydynia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 3 (3)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour invasion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hyperaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Taste disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (10) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin plaque (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral dysaesthesia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Jaundice (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 3 (3)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 4 (4) | 3 (3)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metastases to eye (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Choluria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatocellular injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (6)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (2)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-09-30): https://cdn.clinicaltrials.gov/large-docs/80/NCT02834780/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-07): https://cdn.clinicaltrials.gov/large-docs/80/NCT02834780/SAP_001.pdf